CLINICAL TRIAL: NCT03878199
Title: A Phase I/II, Open-Label, Multi-Center Study Evaluating the Safety and Efficacy of Ruxolitinib and CPX-351 in Combination for the Treatment of Advanced Phase Myeloproliferative Neoplasms
Brief Title: Testing the Effect of Taking Ruxolitinib and CPX-351 in Combination for the Treatment of Advanced Phase Myeloproliferative Neoplasms
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Incyte Corporation (Industry); Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20393; NCI-2019-03712 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Essential Thrombocythemia; Myelofibrosis; Myeloproliferative Neoplasm; Polycythemia Vera; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Thrombocythemia, Essential; Primary Myelofibrosis; Myeloproliferative Disorders; Polycythemia Vera | interventions — Stem Cell Transplantation; CPX-351; Injections; Daunorubicin; Cytarabine; Liposomes; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CPX-351, ruxolitinib, allogeneic SCT) (Experimental): See Detailed Description.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Drug: Ruxolitinib

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic SCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Jakafi; Oral JAK Inhibitor INCB18424

SUMMARY:
This phase I/II trial studies the best dose of ruxolitinib when given together with CPX-351 and to see how well they work in treating patients with accelerated phase or blast phase myeloproliferative neoplasm. Ruxolitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. CPX-351 is a mixture of 2 chemotherapy drugs (daunorubicin and cytarabine) given for leukemia in small fat-based particles (liposomes) to improve the drug getting into cancer cells. Giving ruxolitinib and CPX-351 may work better in treating patients with secondary acute myeloid leukemia compared to CPX-351 alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximum-tolerated dose (MTD) of ruxolitinib in combination with liposome-encapsulated daunorubicin-cytarabine (CPX-351). (Phase I) II. To evaluate the objective response rate in participants with post-myeloproliferative neoplasm (MPN)- accelerated phase (AP)/blast phase (BP) following treatment with the combination of ruxolitinib and CPX-351 (per 2012 MPN-BP criteria). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of ruxolitinib in combination with CPX-351. (Phase I) II. Assess survival outcomes and proportion of patients receiving transplant associated with ruxolitinib in combination with CPX-351. (Phase II)

EXPLORATORY OBJECTIVES:

I. To evaluate the rate of response among participants with MPN-AP/BP using European Leukemia Net (ELN) criteria.

II. Assess the proportion of treated participants with minimal residual disease. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of ruxolitinib followed by a phase II study.

INDUCTION: Patients receive CPX-351 intravenously (IV) over 90 minutes on days 1, 3, and 5 and ruxolitinib orally (PO) twice daily (BID) on days 6-28 of cycle 1.

RE-INDUCTION: Patients with significant residual disease may receive CPX-351 IV on days 1 and 3 and ruxolitinib PO BID on days 4-28 of cycle 2 per the discretion of the treating physician. Patients who have persistent disease following 2 cycles of therapy (induction and re-induction) will be offered salvage chemotherapy.

CONSOLIDATION: Patients that have =< 5% blasts in bone marrow receive CPX-351 IV on days 1 and 3 and ruxolitinib PO BID on days 4-28. Treatment repeats every 28 days for up to 2 cycles provided that counts have partially recovered in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients who successfully complete consolidation therapy with a continued =< 5% blasts in bone marrow and have not undergone an allogeneic stem cell transplantation (SCT) receive ruxolitinib PO BID on days 1-28. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

ALLOGENEIC STEM CELL TRANSPLANTATION: Patients may undergo an allogeneic SCT at any time after achieving =< 5% blasts in bone marrow if they have a suitable donor.

After completion of study treatment, patients are followed up at 30 days and then every 2 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Participants eligible for this study have either MPN in accelerated phase (AP) or blast phase (BP), defined as:

  * MPN-AP is defined by 10% to 19% blasts in the peripheral blood or bone marrow
  * MPN-BP is defined by >= 20% blasts in the blood or bone marrow

    * Either MPN-AP or MPN-BP requires a previous diagnosis of polycythemia vera (PV), essential thrombocythemia (ET), primary or secondary myelofibrosis (MF), or MDS/MPN overlap with intermediate-2 or high risk disease according to IPSS as well as progression on or failure to respond to at least one line of therapy
    * Participants with ET, PV, or MF that have received prior MPN-associated therapy (e.g., hydroxyurea, hypomethylating agents [azacitidine, decitabine], anti-platelet therapies [e.g., aspirin, anagrelide], as well as JAK2 inhibitor therapy [e.g., ruxolitinib or other investigational JAK2 inhibitor]) are eligible. They must discontinue prior to starting therapy; no wash-out is required
* Female participants of childbearing potential must agree to use adequate contraception (2 forms of contraception or abstinence) from the screening visit until 30 days following the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male participants of childbearing potential having intercourse with females of childbearing potential must agree to abstain from heterosexual intercourse or have their partner use 2 forms of contraception from the screening visit until 90 days until the last dose of study treatment. They must also refrain from sperm donation from the screening visit until 90 days following the last dose of study treatment
* Left ventricular ejection fraction at >= 50% as measured by echocardiogram (ECHO) or multigated acquisition (MUGA) scan (14 days prior to initiating study treatment)
* Candidate for cytotoxic-intensive induction chemotherapy
* Willing to take oral medication
* Serum creatinine =< 2 x the upper limit of normal (ULN), or glomerular filtration rate > 20 ml/min/1.73m^2 as calculated by Cockcroft-Gault formula
* Serum potassium, magnesium, and calcium (corrected for albumin) within institutional normal limits or can be corrected with supplementation
* Total serum bilirubin =< 2.5 x ULN
* Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) =< 2.5 x ULN

Exclusion Criteria:

* Ongoing participation in another clinical trial
* Isolated myeloid sarcoma (i.e., participants must have blood or marrow involvement with AML to enter the study)
* Acute promyelocytic leukemia (French-American-British [FAB] M3 classification)
* Active central nervous system (CNS) involvement by AML
* Current treatment or treatment within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of study medication with another investigational medication or current enrollment in another investigational drug protocol (unless there is evidence of rapidly progressive disease in which case a shorter interval from last therapy may be acceptable)
* Any unresolved toxicity equal to or greater than grade 2 from previous anticancer therapy, except for stable chronic toxicities not expected to resolve, such as peripheral neurotoxicity
* Incomplete recovery from any prior surgical procedures or had surgery within 4 weeks prior to study entry, excluding the placement of vascular access
* Disseminated intravascular coagulopathy with active bleeding or signs of thrombosis
* Participants with rapidly progressive disease (defined by blast count doubling within 48 hours) or organ dysfunction that would prevent them from receiving these agents
* Participants with uncontrolled infection will not be enrolled until infection is treated and symptoms controlled

  * Participants with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for >= 72 hours (hrs)
* Known hypersensitivity to ruxolitinib, cytarabine, daunorubicin, or liposomal products
* History of Wilson's disease or other copper metabolism disorder
* Uncontrolled intercurrent illness or any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the participant or compliance with the protocol per investigator's discretion. Including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure, severe uncontrolled ventricular arrhythmias
* Participants with prior cumulative anthracycline exposure of greater than 368 mg/m^2 daunorubicin (or equivalent)
* All participants must discontinue anti-platelet agents or anticoagulants prior to initiation of study drug, including therapeutic doses of aspirin and clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) (Phase I) | Day 1 to day 42
  DLT occurrence after exposure to ruxolitinib and CPX-351.
Proportion of participants that achieve at least an Acute Leukemia Response-Partial response (>= ALR-P, per 2012 myeloproliferative neoplasm - blast phase [MPN-BP] criteria) (Phase 2) | Day 1 to end of induction or re-induction cycle (or upon assessment of the bone marrow biopsy performed near the end of these cycles if this occurs later). Cycle length is 28 days.
  Will compute the proportion of efficacy-evaluable participants achieving overall response rate (ORR) and the exact binominal 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Day 1 to end of 6 cycles with study intervention
  The incidence of treatment-related toxicity and the exact confidence interval will be measured. Each toxicity event will be tabulated and summarized by severity and major organ site according to the CTCAE version (v)5.0.
Incidence of adverse events as assessed by CTCAE version 5.0 | Up to 30 days after last on-study dose
  The incidence of treatment-related toxicity and the exact confidence interval will be measured. Each toxicity event will be tabulated and summarized by severity and major organ site according to the CTCAE v5.0.
Overall survival (OS) | 1 year post treatment
  Time-to-event analysis (e.g., Kaplan-Meier curves or cumulative incidence curves) will be used to evaluate overall survival.
Event-free survival (EFS) | Day 1 to treatment failure, progressive disease, relapse, last exam date, or death (whichever is first), up to 2 years
  Time-to-event analysis (e.g., Kaplan-Meier curves or cumulative incidence curves) will be used to evaluate event-free survival.
Relapse-free survival (RFS) | Date of first documented response (ALR-C) to date of relapse or death from any cause, up to 2 years.
  Time-to-event analysis (e.g., Kaplan-Meier curves or cumulative incidence curves) will be used to evaluate relapse-free survival.
Remission duration | Date of first documented response (ALR-C) to date of documented relapse, up to 2 years
  Time-to-event analysis (e.g., Kaplan-Meier curves or cumulative incidence curves) will be used to evaluate remission duration.
Proportion of participants proceeding to transplant | Date of enrollment to time of transplant or end of follow-up (if no transplant), up to 2 years
  A point estimate and 95% confidence interval will be computed for the proportion of participants who undergo an allogeneic (allo)-SCT (stem cell transplant).

OTHER OUTCOMES:
Proportion of participants that achieve at least a complete remission with incomplete marrow recovery (CRi) (per European Leukemia Net [ELN] criteria) | Day 1 to end of induction or re-induction cycle (up to 8 weeks after start of study treatment)
Rate of CCR; which is the proportion of participants that achieve at least a MLFS (per ELN criteria) | Day 1 to end of induction or re-induction cycle (up to 8 weeks after start of study treatment)
Proportion of participants who have an minimal residual disease (MRD) negative status | End of induction, up to 2 months on study
  Detection of MRD will be achieved by either multi-color flow cytometry (MFC) or next-generation sequencing (NGS) technology and examined using regression based analysis (e.g., logistic regression and Cox regression).
Proportion of participants who have an MRD negative status | End of re-induction, up to 4 months on study
  Detection of MRD will be achieved by either multi-color flow cytometry (MFC) or next-generation sequencing (NGS) technology and examined using regression based analysis (e.g., logistic regression and Cox regression).
Proportion of participants who have an MRD negative status | Up to 12 months on study
  Detection of MRD will be achieved by either multi-color flow cytometry (MFC) or next-generation sequencing (NGS) technology and examined using regression based analysis (e.g., logistic regression and Cox regression).
Frequency of each mutation (single nucleotide polymorphism [SNP]) | End of induction or re-induction, up to 2 months on study

CONTACTS AND LOCATIONS:
Overall Officials: Uma Borate, MD, Principal Investigator — The Ohio State Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OHSU, Portland, Oregon
  - Simmons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu